CLINICAL TRIAL: NCT05015933
Title: Feasibility, Safety and Effectiveness of Intrathecal Pump Refills at Home: a Pilot Study.
Brief Title: Intrathecal Pump Refills at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCAPE
Record Dates: First submitted 2021-08-02; First posted 2021-08-23 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Intrathecal Drug Delivery; Implantable Pump; Telemedicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refill at home (Experimental): Patients will have one pump refill at home instead of at the hospital.
  Interventions: Procedure: Pump refill procedure at home

INTERVENTIONS:
Procedure: Pump refill procedure at home — Implantable pump refill is performed at home

SUMMARY:
The aim of this pilot study is to evaluate the feasibility, safety and effectiveness of intrathecal pump refill procedures at home. It is our hypothesis that a refill at home will be safe, effectiveness and feasible, as is demonstrated in The Netherlands, and preferred by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient receives intrathecal drug therapy
* Patient is at least 18 years old
* Native French-or Dutch speaking persons.

Exclusion Criteria:

* Patients < 18 years old.
* No native Dutch or French speaking persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Once, at the moment of the study visit, immediately after the pump refill
  A seven-point Likert scale asking the patient to rate the overall level of satisfaction with the refill at home will be used.
Successful pump refill | Once, at the moment of the study visit, immediately after the pump refill
  A binary variable to indicate success or failure of this intervention, reported by the physician.
Patient safety | Once, at the moment of the study visit, immediately after the pump refill
  A seven-point Likert scale asking the patient to rate the overall level of safety with the refill at home will be used.
Physician safety | Once, at the moment of the study visit, immediately after the pump refill
  A seven-point Likert scale asking the physician to rate the overall level of safety with the refill at home will be used.

SECONDARY OUTCOMES:
Environmental safety | Once, at the moment of the study visit, immediately after the pump refill
  An open question in which the physician can indicate whether there were any situations that were not safe.
Clean, sterile procedure | Once, at the moment of the study visit, immediately after the pump refill
  An open question in which the physician can mention all potential risks.
An objective confirmation of correct injection in the pump by ultrasound. | Once, at the moment of the study visit, immediately after the pump refill
  After the refill procedure is performed, an ultrasound will be made to visually ensure that the refill was correctly performed without loss of liquor outside the pump.
Adverse events | Once, at the moment of the study visit, immediately after the pump refill
  All adverse events will systematically be reported by the physician.
Patient feasibility | Once, at the moment of the study visit, immediately after the pump refill
  A seven-point Likert scale asking the patient to rate the overall level of feasibility with the refill at home will be used.
Quality of teleconsultant connection by teleconsultant | Once, at the moment of the study visit, immediately after the pump refill
  Quality of the internet connection will be evaluated by the teleconsultant.
Time burden for teleconsultant | Once, at the moment of the study visit, immediately after the pump refill
  The time will be measured from the beginning until the end of the call.
Physician feasibility | Once, at the moment of the study visit, immediately after the pump refill
  A seven-point Likert scale asking the physician to rate the overall level of feasibility with the refill at home will be used.
Quality of teleconsultant connection by physician | Once, at the moment of the study visit, immediately after the pump refill
  Quality of the internet connection will be evaluated by the physician.
Time burden for physician | Once, at the moment of the study visit, immediately after the pump refill
  The time will be measured from the beginning until the end of the call.
Patient preference | Once, at the moment of the study visit, immediately after the pump refill
  Patients will be asked to indicate whether they prefer to have their next refill at home.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium